CLINICAL TRIAL: NCT03159403
Title: Retrospective, Observational Evaluation of the Utilization, Outcomes, and Adverse Events Associated With Orbactiv® for the Treatment of Infections Presumed or Confirmed to be Caused by Gram Positive Bacteria in a Real World Setting
Brief Title: A Retrospective Observational Study to Evaluate the Utilization, Outcomes, and Adverse Events in Participants Treated With Orbactiv® (Oritavancin) for Infections Caused by Gram Positive Bacteria in a Real World Setting
Status: Completed | Type: Observational
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDCO-ORI-15-05
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Gram-Positive Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — oritavancin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oritavancin: Participants who received at least one dose (at least one for 3 hours per dose) of oritavancin intravenous (IV) as monotherapy or part of a broader regimen. The maximum number of doses to be received by a participant is not known at this time.
  Interventions: Drug: Oritavancin

INTERVENTIONS:
Drug: Oritavancin — This study is an observational study. All participants were administered oritavancin prior to enrollment in this study.
  Other Names: Orbactiv®

SUMMARY:
This study is a retrospective, observational study to evaluate oritavancin use in participants under real world conditions.

ELIGIBILITY:
Inclusion Criteria:

* The participant was treated with at least one dose of oritavancin for a suspected or confirmed gram positive infection, as monotherapy or part of a broader regimen.
* At least 60 days has elapsed since the participant received the last dose of oritavancin therapy (prior to data entry into the electronic Case Report Form).

Exclusion Criteria:

* The participant received oritavancin as a part of a controlled clinical trial.
* The participant received oritavancin as a part of a Medicines Company-sponsored single or multi-centered pharmacoeconomic outcomes study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in real world settings (which include infusion centers, clinics, emergency departments, and observation and inpatient hospital beds), who received at least one dose of oritavancin.
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Types Of Primary Infections Being Treated With Oritavancin | Day 1
  The Types Of Primary Infections refers to whether the primary infection was skin or skin structure or other systemic infection (for example, bacteremia, prosthetic joint infection, osteomyelitis).
Classification Of Primary Infections Being Treated With Oritavancin | Day 1
  The classification of primary infection refers to whether a skin or skin structure infection was cellulitis, abscess, wound, or other.
Proportion Of Participants With Positive Cultures For Gram Positive, Gram Negative, And Anaerobic Pathogens From The Infected Site | Up to 30 days after oritavancin IV infusion
  All microbiology results during the infection event will be reported. Microbiology results will be noted only for the infection site for which oritavancin (in addition to other agents) is administered or other site related to the primary infection in case of multiple infections. An adverse event was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.
Duration Of Treatment With Oritavancin | Day 1 through end of oritavancin IV infusion
  The number of days of treatment with oritavancin will be presented.
Proportion Of Participants With A Clinical Outcome Of Cure, Improved, or Failure | Up to 30 days after oritavancin IV infusion
  Clinical assessments will be based on participant records between end of infusion to 30 days following the last dose of Oritavancin. Clinical categories for assessment include:
  * Cure - Clinical signs and symptoms are resolved, and no additional antibiotic therapy is necessary for the treatment of the infection
  * Improved - Partial resolution of clinical signs and symptoms, and no additional antibiotic therapy is necessary for the treatment of the infection
  * Failure - Inadequate resolution, or new or worsening clinical signs and symptoms, such that additional antibiotic therapy is necessary for treatment of the infection
  * Non-evaluable - Unable to determine response because the participant record did not contain the necessary information to determine cure, improvement, or failure
Proportion Of Participants With A Microbiologic Eradication Or Microbiologic Persistence | Up to 30 days after oritavancin IV infusion
  Microbiological assessments will be based on participant records between end of infusion to 30 days following the last dose of oritavancin. Microbiological categories will include only gram positive pathogens believed to be related to the infection process and are defined as:
  * Microbiologic eradication (the baseline gram positive pathogen has been eradicated)
  * Microbiologic persistence (the baseline gram positive pathogen persists)
  * Culture drawn post-oritavancin therapy, but no information regarding microbiologic culture results
  * No culture collected following the last dose of oritavancin
  * No information available
Use Of Concomitant Antibiotics With Oritavancin | Day 1 through end of oritavancin IV infusion
  Concomitant antibiotics include those used between the first and last dose of oritavancin. The number of participants and the type of antibiotic taken will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Global Health Science Center
Locations (21):
- United States (21):
  - Birmingham Infectious Disease and Infusion, Birmingham, Alabama
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Florida Infectious Disease Care, Fort Myers, Florida
  - Infectious Diseases Associates of North Central Florida, LLC, Ocala, Florida
  - WellStar Health System - Kennestone, Marietta, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - St. Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - IDC Clinical Research, LLC, Wichita, Kansas
  - Clinical Infectious Disease Specialists, Las Vegas, Nevada
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Erie County Medical Center, Buffalo, New York
  - Trinity Health Medical Group, Minot, North Dakota
  - Infectious Diseases Consultants of OKC, Oklahoma City, Oklahoma
  - TruCare Internal Medicine and Infectious Diseases, DuBois, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Center for Infectious Diseases & Travel Medicine, El Paso, Texas
  - Houston Center For Infectious Diseases, The Woodlands, Texas
  - Infectious Disease and Pulmonary, Victoria, Texas
  - Foot & Ankle Institute, St. George, Utah

IPD SHARING:
Plan to Share IPD: No